CLINICAL TRIAL: NCT03393195
Title: Study of Time-restricted Eating on Weight Loss. A Randomized Controlled Trial of the Effects of Time-restricted Eating on Weight Loss in Obese Subjects.
Brief Title: Study of Time-restricted Eating on Weight Loss.
Acronym: TREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-22110
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: Weight loss; Diet; Time-restricted feeding
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Loss; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. Participants will randomly assigned to one of two diet interventions for the duration of the 12-week study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating plan (Experimental): Participants in this group will be instructed to fast every day from 8pm until 12pm the following day. From 12pm until 8pm, participants can eat and drink whatever they want. During fasting hours, participants can drink water and black coffee.
  Interventions: Behavioral: Time-restricted Eating plan
- Consistent Meal Timing Plan (Active Comparator): Participants in this group will be instructed to eat three daily meals during specified eating times. Their first meal will be between 7am-11am. Second meal between 11am and 3pm, and third meal between 4pm-10pm. Participants will be encouraged to eat small snacks if needed so that they can eat their next meal during the specified window.
  Interventions: Behavioral: Consistent Meal timing plan

INTERVENTIONS:
Behavioral: Time-restricted Eating plan — Research team will prescribe an eating plan for the participant to follow for the 12 week study. The eating plan will consist of eating during a specified 8 hour window and fasting for the remaining 16 hours of the day.
  Arms: Time-restricted eating plan
Behavioral: Consistent Meal timing plan — Research team will prescribe an eating plan for the participant to follow for the 12 week study.The eating plan will consist of eating three structured meals each day during three specified meal windows.
  Arms: Consistent Meal Timing Plan

SUMMARY:
This is a randomized controlled trial studying the effects of time-restricted eating (TRE) on weight loss in obese humans. Obesity is the number one risk factor for type 2 Diabetes Mellitus (T2DM), and numerous studies demonstrate that weight loss is an effective strategy to prevent T2DM and improve the metabolic health of people diagnosed with T2DM. Unfortunately, classical calorie restriction diets often fail to produce long-term weight loss due to low compliance, reduced resting metabolic rate (RMR), and other factors. Therefore, novel dieting techniques must be explored in order to successfully treat obesity and prevent T2DM. Studies in mice provide compelling evidence that feeding/fasting cycles can be altered to produce beneficial effects on weight loss and metabolic health markers in the absence of calorie restriction. Limited research in human subjects suggests that this feeding paradigm may translate to human health as well, however, more research needs to be done in order to confirm this hypothesis. This study will determine if TRE can lead to weight loss in obese human subjects. Secondary outcomes include changes in body composition, HOMA-IR, hormonal and biochemical serum markers, RMR, and total energy expenditure (TEE).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-40 kg/m2
* Participants must regularly consume breakfast (at least 5 days per week)
* Must speak, read, and comprehend English
* Access to reliable internet and/or wifi
* Must have a valid email address and phone number
* Must have a cellular phone with data plan

Exclusion Criteria:

* HIV or immunocompromised
* Current or past cancer diagnosis
* Pregnant, breastfeeding, or planned pregnancy in next 6 months
* Beginning or ending hormonal contraception in next 6 months
* Current diagnosis of type or type 2 diabetes
* Currently taking glucose-lowering drugs, statins, or oral steroids
* History of gastric bypass surgery or any other weight-loss surgery
* History of anorexia or bulimia
* Frequent travel across time zones or unusual work hours
* Unable to fast for prolonged periods due to medical condition
* Unable to stand for several minutes without aid
* Cannot lie down on cushioned table for 30 minutes
* No internal metal artifacts that would alter body composition
* Unable to travel to UCSF for in-person testing
* Requires translator services

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Weight Loss | Daily for 12 weeks
  Measure changes in weight during the 12 week study

SECONDARY OUTCOMES:
Fat loss | Measured twice: Once at study start and once 12 weeks later
  Measure changes in fat mass during the 12 week study using DXA data
Changes in lean mass | Measured twice: Once at study start and once 12 weeks later
  Measure changes in lean mass during the 12 week study using DXA data
Fasting insulin levels | Measured twice: Once at study start and once 12 weeks later
  Measure fasting insulin levels pre and post intervention
Resting metabolic rate | Measured twice: Once at study start and once 12 weeks later
  Will measure participants resting metabolic rate
Total energy expenditure | Measured twice: Once at study start and once 12 weeks later
  Will measure participants total energy expenditure during the week leading up to the study start and during the final week of the study
Changes in fasting glucose levels | Measured twice: Once at study start and once 12 weeks later
  WIll measure fasting blood glucose levels prior to diet intervention and again at study completion
Changes in HbA1c levels | Measured twice: Once at study start and once 12 weeks later
  WIll measure HbA1c levels prior to diet intervention and again at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Ethan J Weiss, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong MC, Bennett JP, Leong LT, Tian IY, Liu YE, Kelly NN, McCarthy C, Wong JMW, Ebbeling CB, Ludwig DS, Irving BA, Scott MC, Stampley J, Davis B, Johannsen N, Matthews R, Vincellette C, Garber AK, Maskarinec G, Weiss E, Rood J, Varanoske AN, Pasiakos SM, Heymsfield SB, Shepherd JA. Monitoring body composition change for intervention studies with advancing 3D optical imaging technology in comparison to dual-energy X-ray absorptiometry. Am J Clin Nutr. 2023 Apr;117(4):802-813. doi: 10.1016/j.ajcnut.2023.02.006. Epub 2023 Feb 14. PMID 36796647
- [Derived] Lowe DA, Wu N, Rohdin-Bibby L, Moore AH, Kelly N, Liu YE, Philip E, Vittinghoff E, Heymsfield SB, Olgin JE, Shepherd JA, Weiss EJ. Effects of Time-Restricted Eating on Weight Loss and Other Metabolic Parameters in Women and Men With Overweight and Obesity: The TREAT Randomized Clinical Trial. JAMA Intern Med. 2020 Nov 1;180(11):1491-1499. doi: 10.1001/jamainternmed.2020.4153. PMID 32986097

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03393195/Prot_SAP_000.pdf